CLINICAL TRIAL: NCT01182480
Title: Chronic Care Management/Patient Relationship Management Proof of Concept
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Microsoft Corporation (Industry); EMC Consulting (Unknown)
Responsible Party: Principal Investigator, Andrew W. Steele, MD, MPH, MSc, Director, Medical Informatics, Denver Health and Hospital Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: COMIRB 10-0257
Record Dates: First submitted 2010-08-11; First posted 2010-08-16 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Patient Relationship Management (PRM) Program — Patients will be contacted through SMS text messaging under the following circumstances:
  * 7 days, 2 days, and 1 day before scheduled appointments. Messages will contain the date, time, and location where the appointment is scheduled. Patients will be prompted to respond with 'YES' if they are able to keep their appointment, and 'NO' if they need to reschedule. An acknowledgement of receipt will be sent in response to all patient-initiated messages.
  * 3 days per week to request that patients respond with fasting blood sugar measurements. An acknowledgement of receipt will be sent in response to all patient-initiated messages.

SUMMARY:
This proof of concept study proposes to evaluate the feasibility of a communications-technology-based chronic care and patient relationship management program to improve diabetes self management among adult diabetic patients in an urban safety net population by providing between-visit reminders and chronic disease support through cell phone text messaging.

The investigators hypothesize that diabetic patients enrolled in the program will be less likely to miss scheduled appointments and will have greater perceived self-efficacy and improved patient satisfaction concerning chronic disease management. No-show rates among patients enrolled in the program are expected to be lower than among patients receiving standard care.

ELIGIBILITY:
Inclusion Criteria:

* patients with diabetes
* receive care at a primary care clinic in the DH system
* between 18 and 76 years of age
* primary language of English or Spanish
* ownership of a qualifying cell phone (SMS text capable)
* ownership of a glucometer.

Exclusion Criteria:

* life expectancy less than six months,
* do not have or cannot use a phone or glucometer
* do not want to participate

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Steele, MD, MPH, Principal Investigator — Denver Health and Hospital Authority
Locations (1):
- Denver Health and Hospital Authority, Denver, Colorado, United States

REFERENCES:
- [Result] Fischer HH, Moore SL, Ginosar D, Davidson AJ, Rice-Peterson CM, Durfee MJ, MacKenzie TD, Estacio RO, Steele AW. Care by cell phone: text messaging for chronic disease management. Am J Manag Care. 2012 Feb 1;18(2):e42-7. PMID 22435883

RESULTS

PARTICIPANT FLOW:
Recruitment Details: English and Spanish-speaking adult patients (18-76 years old) with diabetes in possession of cell phones who receive primary care at Sam Sandos Westside Family Health Center (Westside), a federally qualified community health center in the Denver Health integrated healthcare system in Denver, CO.
Pre-assignment Details: Exclusion criteria included a life expectancy less than six months, age < 18 or > 76, and either lacking possession of or inability to use a cell phone or glucometer.
Groups:
- Text Intervention: Group of study participants who received the text message intervention over a 3-month period. Participants received text messages 7, 2, and 1 day(s) prior to each of their scheduled appointments as recorded in the Denver Health scheduling system, and also received text messages prompts 3 times per week asking them to provide fasting blood sugar readings.
Period: Overall Study
Arm/Group | Text Intervention
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Text Intervention: Group of study participants who received the text message intervention over a 3-month period.
Arm/Group | Text Intervention
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.29 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Patient Engagement
Description: Patient engagement was assessed by patient text message response rates and average response times. Response rates were calculated as a percentage from the number of patient-initiated text messages sent in response to a system-generated request for information (the numerator) divided by the total number of system-generated requests for information (the denominator). Average response times were calculated from system-recorded time stamps for outbound requests sent and inbound patient-initiated responses received.
Time Frame: 3 months
Population: Group of study participants who received the text message intervention over a 3-month period.
Measure: Number; unit: text message response rate (percent)
Arm/Group | Text Intervention
Number analyzed (Participants) | 47
text message response rate (percent) | 68.14

2. Secondary Outcome: Appointment Attendance
Description: As measured by no-show rates for appointments at all clinics during the study period, compared between intervention and control groups
Time Frame: 3 months
Reporting Status: Not Posted

3. Secondary Outcome: Perceived Self-efficacy
Description: As measured by comparison of patient responses to validated assessment instrument administered at baseline and post-intervention
Time Frame: 3 months
Reporting Status: Not Posted

4. Secondary Outcome: Glycemic Control
Description: Measured by patients' self-reported fasting blood glucose levels during the intervention period and compared to previous laboratory data in the medical record.
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Text Intervention
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

LIMITATIONS AND CAVEATS:
Insufficient power (# appointments) to detect changes in attendance rates; technical issues with self-efficacy data resulting in inability to compare pre- and post- intervention; intervention period insufficient to assess impact on glycemic control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes